CLINICAL TRIAL: NCT05501002
Title: US Pilot Study to Evaluate the Safety and Effectiveness of the CereVasc® EShunt® System in the Treatment of Communicating Hydrocephalus
Brief Title: Pilot Study to Evaluate the CereVasc® EShunt® System in the Treatment of Communicating Hydrocephalus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: CereVasc Inc (Industry)
Collaborators: AlvaMed, Inc. (Industry); Simplified Clinical Data Systems, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0029
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Hydrocephalus; Hydrocephalus, Communicating
Keywords: eShunt; Endovascular Shunt
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device Arm (Experimental): The Device Arm receives the eShunt® Implant
  Interventions: Device: eShunt® Implant

INTERVENTIONS:
Device: eShunt® Implant — The eShunt® Implant is intended to drain excess cerebrospinal fluid from the intracranial subarachnoid space to the venous system as a less invasive therapy for treating hydrocephalus.
  Other Names: eShunt®; eShunt® system

SUMMARY:
The purpose of this study will be to evaluate a novel, minimally invasive method of treating hydrocephalus in adults. The eShunt® System includes a proprietary eShunt® Delivery System and the eShunt® Implant, a permanent implant that is deployed in a mildly invasive, neuro-interventional procedure. The eShunt® Implant is designed to drain excess cerebrospinal fluid (CSF) from the intracranial subarachnoid space (SAS) into the venous system.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open label, pilot study of the eShunt® System. The study population consists of patients with post-aneurysmal subarachnoid hemorrhage (SAH) treated for increased intracranial pressure (ICP) resulting in symptomatic hydrocephalus using an external ventricular drain (EVD) to facilitate CSF drainage and who cannot be "weaned" from the EVD after the hemorrhagic event.

After completion of the procedure to place the eShunt® device, the ICP will be monitored and recorded for up to 48 hours. Subjects will then return for follow-up visits that include standard neurological evaluations at 30, 60, 90, 180, and 365 days postimplantation; imaging will also be acquired at 30, 90 and 365 days after implant. Subjects will continue to attend follow-up visits every 180 days thereafter until the study is closed or up to 5 years post-implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 21 years old
* Patient or legally authorized representative is able and willing to provide written informed consent
* Post-aneurysmal SAH with Hunt and Hess Grades I-IV with EVD in place for at least 7 days with the need for a permanent CSF shunt determined through a failed EVD clamping trial defined as:

  1. Post-clamping ICP of > 20 cmH2O for 15 minutes, or
  2. Post-clamping ICP > 25 cmH2O for < 15 minutes with patient intolerance to EVD clamping, or
  3. Significant radiographic signs of increasing ventriculomegaly, or
  4. Neurological decline attributable to ventriculomegaly and requiring CSF diversion
* Clinical signs and symptoms of communicating hydrocephalus
* Neurologically stable without evidence of severe vasospasm
* Pre-procedure MRI confirmation of anatomy suitable for eShunt Procedure, as described in Section 1.8.3.4.2 and confirmed by subject screening committee (SSC)
* Pre-procedure CT confirmation of anatomy suitable for eShunt Procedure, as described in Section 1.8.3.4.2 and confirmed by SSC

Exclusion Criteria:

* Presence of gross blood in CSF
* Signs or symptoms of obstructive hydrocephalus
* Active systemic infection or infection detected in CSF
* Prior or existing shunts, endoscopic third ventriculostomy, or any previous surgical intervention for hydrocephalus
* Hypersensitivity or contraindication to heparin or radiographic contrast agents which cannot be adequately pre-medicated, desensitized or where no alternative is available
* Occlusion or stenosis of the internal jugular vein
* Venous distension in the neck on physical exam
* Medical conditions associated with prolonged elevation of jugular venous pressure, including jugular vein stenosis or stricture, right sided heart failure, cirrhosis of the liver, arterial venous fistulas in the arm for dialysis purposes, or an arterial venous fistula or malformation in the neck or brain
* Atrial septal defect or patent foramen ovale identified on cardiac echocardiogram
* History of bleeding diatheses, coagulopathy or will refuse blood transfusion in cases of emergency
* Stroke or transient ischemic attack within 180 days of eShunt Procedure
* Presence of a deep vein thrombosis superior to the popliteal vein
* International Normalized Ratio (INR) or Partial Thromboplastin Time (PTT) results outside of normal range (INR 0.8-1.4; PTT 25-35 seconds)
* Presence of a posterior fossa tumor or mass
* Life expectancy < 1 year
* Currently participating in another investigational drug or device trial that could conflict with study data collection or follow-up
* Pregnant
* Unwilling or unable to comply with follow-up requirements

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Reduction in ICP | 24-48 hours after eShunt Implant placement
  At 24 to 48 hours after eShunt Implant deployment (with EVD remaining clamped) an ICP measurement that indicates:
  * ICP below 20 cmH2O with no periods longer than 15 minutes above 20 cmH2O
  * No episodes of ICP above 25 cmH2O with associated symptoms

SECONDARY OUTCOMES:
Occurrence of Serious Adverse Events | 90 days post procedure
  The number of device and/or procedure-related serious adverse events (SAEs) after the implant procedure will be calculated.
Incidence of clinically significant changes in Computed Tomography Imaging (CT/CTA) from baseline. | 1 year post procedure
  Clinically significant changes from baseline CT images will be summarized
Number of participants with clinically significant changes in physical and neurologic examination assessments from baseline | 1 year post procedure
  Clinically significant changes from baseline physical examination and neurologic examination assessments will be summarized
Summary of Adverse Events | 90 days post procedure and at study completion
  Tabulation of all Adverse Events collected in the study.
Changes in Modified Rankin Scale Scores | 1 year post procedure
  Changes in Modified Rankin Scale scores from baseline will be summarized.
Number of subjects requiring conversion to conventional CSF shunt | 1 year post procedure
  Evaluate the need for CSF diversion by conventional CSF shunt insertion within 12 months after eShunt Implant deployment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Montefiore Medical Center Department of Neurosurgery, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lylyk P, Lylyk I, Bleise C, Scrivano E, Lylyk PN, Beneduce B, Heilman CB, Malek AM. First-in-human endovascular treatment of hydrocephalus with a miniature biomimetic transdural shunt. J Neurointerv Surg. 2022 May;14(5):495-9. doi: 10.1136/neurintsurg-2021-018136. Epub 2021 Dec 3. PMID 34862267
- [Background] Heilman CB, Basil GW, Beneduce BM, Malek AM. Anatomical characterization of the inferior petrosal sinus and adjacent cerebellopontine angle cistern for development of an endovascular transdural cerebrospinal fluid shunt. J Neurointerv Surg. 2019 Jun;11(6):598-602. doi: 10.1136/neurintsurg-2018-014445. Epub 2019 Jan 9. PMID 30626626